CLINICAL TRIAL: NCT06700200
Title: The Effect of Non-invasive Transauricular Vagus Nerve Stimulation on Upper Gastrointestinal Motility in Healthy Individuals
Brief Title: TVNS and Upper GI Motility
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Other
Other Study IDs: NL86446.068.24
Record Dates: First submitted 2024-10-23; First posted 2024-11-21 (Actual); Last update posted 2024-11-21 (Actual); Status verified 2024-11

CONDITIONS: Healthy Volunteer

STUDY DESIGN:
Intervention Model Description: Subjects will receive two types of stimulation (i.e. taVNS vs sham) during a measurement with an antroduodenal manometry. The order of stimulation applied during each block is randomized.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Participant and investigator will not know the randomization order of tVNS
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- taVNS (Active Comparator): The vagus nerve will be stimulated transcutaneously. The concha of the left ear will be stimulated.
  Interventions: Device: taVNS
- Sham stimulation (Placebo Comparator): The vagus nerve will be stimulated transcutaneously. The concha of the left ear will be stimulated. The device is inactive.
  Interventions: Device: taVNS

INTERVENTIONS:
Device: taVNS — transauricular vagus nerve stimulation

SUMMARY:
To study the impact of tVNS on gut motor function, with regards to its potential to induce phase III contractions in the upper GI tract, in healthy subjects.

Hypothesis: We hypothesize that tVNS will induce on average an excess of 1 additional phase III contraction of antral origin in the fasted period compared to sham stimulation.

DETAILED DESCRIPTION:
Healthy volunteers (n=12) will be recruited, both male and female, aged aged 18-55 years old. Participants will arrive after an overnight fast at the GI physiology unit ('functiekamer') of the Maastricht University Medical Center, where they will be inserted an antroduodenal manometry catheter through the nose into the duodenum under fluoroscopy control. The high-resolution catheter contains 36 transducers spaced at 1-cm intervals (Unisensor AG, Attikon, Switzerland). Using this catheter, stomach and duodenum motility patterns will be recorded for 8 hours.

Participants will undergo tVNS (cymba concha of the left ear) alternated with sham (a non-conducting electrode) in a blinded pre-randomized fashion using 2 blocks of 4 hours during the 8-hour registration period. In addition, blood samples will be taken at baseline and at intervals of 30 minutes during the 8-hour test period. Levels of the GI hormones motilin and PP will be measured as surrogate markers of vagal efferent influence on GI motor function.

Autonomic parameters will be registered using pulse plethysmography. A wearable device (Shimmer3 GSR Sensor) will also be used to measure heart rate variability and skin conductance. Heart rate variability is regarded as a parameter reflecting cardiac parasympathetic activity.(33, 34) The root mean square of successive differences (RMSSD) is a commonly utilized and thoroughly validated measure of heart (and pulse) rate variability. (35, 36).

After the 8-hour registration period, all measurement equipment and the iv. cannula is removed. Participants are provided a meal voucher to be consumed at the hospital visitor's restaurant, whereafter the test day is finished.

ELIGIBILITY:
Inclusion Criteria:

* Healthy participants (defined as those without a pre-existing medical comorbidity, including those without a history of cardiac arrhythmia).
* Age between 18 and 55 years.
* Ability to understand and speak the Dutch language.

Exclusion Criteria:

* Pregnancy or lactation.
* Use of any substances (such as medication or recreational drugs) influencing gastrointestinal motility
* Not meeting the inclusion criteria above.
* Students and employees of Maastricht University are not precluded from participation, unless they have a direct personal, professional of hierarchical position with regards to any of the study team members or their department.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Estimated)
Dates: Start 2024-12-01 (Estimated); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Phase III Antral contractions | During ADM
  A clinically meaningful increase in the number of phase III contractions of antral origin in the fasted period during the tVNS stimulation compared to the sham stimulation.

SECONDARY OUTCOMES:
Motilin and pancreatic polypeptide levels | During ADM
  Blood samples will be taken every 30 minutes
Other ADM parameters | During ADM
  * Antral and duodenal contraction frequency,
  * Contraction amplitude,
  * Motility index: MI=ln((contractionfrequency∗amplitude)+1),
  * Number of duodenal phase II contractions
  * Number of MMCs.

CONTACTS AND LOCATIONS:
Overall Officials: D Keszthelyi, Principal Investigator — Maastricht UMC

IPD SHARING:
Plan to Share IPD: No